CLINICAL TRIAL: NCT05137041
Title: A Phase IIIB Randomized, Open Label, Two Arms and Parallel Group Clinical Trial to Assess the Efficacy and Safety of FIRTECH (Infrared Therapy Patch), for Treating Patients Suffering From Mild to Moderate Acute Low Back Pain
Brief Title: Efficacy and Safety of FIRTECH in Patients With Mild to Moderate Acute Low Back Pain
Acronym: IRPATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS16453; U1111-1255-4648 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-11-18; First posted 2021-11-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITP FIRTECH (Experimental): The ITP FIRTECH patch was applied on the lower back region of the body on Day 1 and intended to be worn for 5 Days (Day 5).
  Interventions: Device: ITP FIRTECH
- No Patch Control Arm (No Intervention): No patch application.

INTERVENTIONS:
Device: ITP FIRTECH — Infrared Therapy Patch
  Arms: ITP FIRTECH

SUMMARY:
Primary Objective:

To assess the efficacy of the infrared therapy patch (ITP) FIRTECH for treating participants suffering from mild to moderate acute low back pain.

Secondary Objectives:

* To assess the efficacy of ITP FIRTECH on participant disability
* To assess the efficacy of ITP FIRTECH on the degree of participant mobility
* To assess the safety of ITP FIRTECH

DETAILED DESCRIPTION:
Duration of study participation is up to 6 days per participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from mild to moderate acute low back pain
* Low back pain (lumbar back pain) is defined as pain in the back from the level of the lowest rib down to the gluteal fold
* Acute episode is defined as acute pain with less than 1 month duration
* With intensity less than or equal to 6 on 0-10 Numerical Rating Scale (NRS)

Exclusion Criteria:

* Participants suffering from any neurological pathology which could be responsible of the pain
* Participants suffering from leg pain irradiation
* Participants suffering from chronic lumbar pain of any etiology
* Participants with chronic arthrosis and neurological symptoms
* Participants experiencing recent significant trauma (i.e., injury related to a fall from a height or motor vehicle crash, or from a minor fall or heavy lifting in a participants with osteoporosis or possible osteoporosis)
* Participants with major or progressive motor or sensory deficit, new-onset bowel or bladder incontinence or urinary retention, loss of anal sphincter tone, saddle anesthesia, history of cancer metastatic to bone, and suspected spinal infection
* Participants clinically diagnosed with anxiety and/or depression
* Participants using any medication for their pain within the last 48 hours within enrollment into the study
* Participants taking any systemic medication for their pain within the last 24 hours (48 hours for diclofenac or corticosteroids)
* Participants currently using recreational or illicit drugs or with a recent history of drug or alcohol abuse or dependence
* Participants with any other medical condition that would interfere with efficacy and safety assessments based on investigator's judgment
* Participants having received non-pharmaceutical lower back pain treatment (physiotherapy, heat treatment or massage) within 12 hours prior to enrollment
* Participants having received spinal injection back pain treatment within 6 months prior to enrollment
* Participants having received surgery due to back pain or rehabilitation due to back pain in the last 12 months
* Participants with a known sensitivity to paracetamol
* Participants with known cutaneous hypersensitivity to plaster
* Participants participating in another clinical study within the past 30 days
* Participants who are pregnant or breastfeeding; contraception is mandatory
* Participants having damaged, non-intact, or scarred skin in or near the point of patch application
* Participants having a known skin sensitivity
* Participants having impaired blood circulation

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Germany (4):
  - Investigational Site Number :06, Bad Homburg
  - Investigational Site Number :02, Leipzig
  - Investigational Site Number :01, Munich
  - Investigational Site Number :03, Weinheim
- Italy (3):
  - Investigational Site Number :7, Taormina, Messina
  - Investigational Site Number :5, Alessandria
  - Investigational Site Number :4, Chieti

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16453 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25281&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 221 participants took part in the study at 7 investigative sites in Germany and Italy from 04 November 2021 to 22 November 2022.
Pre-assignment Details: Participants suffering from mild to moderate acute low back pain were randomly assigned in a 1:1 ratio to receive either FIRTECH patch or no patch.
Groups:
- ITP FIRTECH: The infrared therapy patch (ITP) FIRTECH patch was applied on the lower back region of the body on Day 1 and intended to be worn for 5 Days (Day 5).
Period: Overall Study
Arm/Group | ITP FIRTECH | No Patch Control Arm
Started | 113 | 108
Intent-to-Treat Population (Intent-to-Treat population was defined as all participants randomized.) | 113 | 108
Safety Population (Safety population was defined as all participants randomized into the study and, if randomized to the "patch" arm, had the device installed.) | 114 (The Safety Population included a participant that was randomized to the no patch arm of the study, but did receive the FIRTECH Patch.) | 107 (The Safety Population included a participant that was randomized to the no patch arm of the study, but did receive the FIRTECH Patch.)
Modified Intent-to-Treat Population (Modified Intent-to-Treat population was defined as all participants randomized that had the Numerical Rating Scale (NRS) evaluation done at baseline and Day 5 with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0").) | 91 | 89
Full Analysis Set (Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0").) | 97 | 84
Completed | 112 | 104
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population was defined as all participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | ITP FIRTECH | No Patch Control Arm | Total
Number analyzed (Participants) | 113 | 108 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.10) | 44.7 (12.87) | 45.2 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
  Male | 54 | 46 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Numerical Rating Scale (NRS) Responders at Day 5
Description: NRS is used to assess pain intensity, it is a 11-point scale (0-10) where '0' representing 'no pain' and '10' representing 'worst pain imaginable'. Responder is defined as participant with ≥30% decrease from baseline in pain NRS and who did not take rescue medication (defined as receiving paracetamol (authorized), any other analgesics and anti-inflammatory drugs as well as any non-pharmaceutical therapy (prohibited) for treating pain starting from randomization to Day 5 or starting before the study and still ongoing at randomization).
Time Frame: Day 5
Population: Modified Intent-to-Treat population was defined as all participants randomized that had the Numerical Rating Scale (NRS) evaluation done at baseline and Day 5 with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0").
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 91 | 89
percentage of participants | 72.5 [62.17 to 81.37] | 49.4 [38.67 to 60.25]
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.002, Fisher Exact

2. Secondary Outcome: Number of Participants Reported With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A treatment emergent adverse event (TEAE) is an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.
Time Frame: Day 1 to Day 6
Population: Safety population was defined as all participants randomized into the study and, if randomized to the "patch" arm, had the device installed.
Measure: Count of Participants; unit: Participants
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 114 | 107
Participants | 18 | 7

3. Secondary Outcome: Normalized Sum of Pain Intensity Difference (PID) Over 5 Days (SPID0-5)
Description: NRS is used to assess pain intensity, it is a 11-point scale (0-10) where '0' representing 'no pain' and '10' representing 'worst pain imaginable'. PID equals the NRS change from baseline. A negative difference indicates improvement. Time-weighted summed pain intensity difference (SPID) was calculated by multiplying the PID score at each postdose time point by the duration since the preceding time point and then summing these values. The Normalized Sum of Pain Intensity Difference (SPID0- 5) is to be calculated as the SPID0- 5 divided by the total duration time. The score range for ITP FIRTECH arm is -5.0 to 2.1 and for no patch control arm is -5.8 to 3.1.
Time Frame: Baseline, Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0").
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
units on a scale | -1.52 (1.356) | -0.91 (1.484)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.015, ANCOVA; The p-value was adjusted using a False Discovery Rate approach (Benjamini-Hochberg); Least Square Mean Difference = -0.5, 95% CI 2-sided [-0.817 to -0.137], Standard Error of Mean 0.17

4. Secondary Outcome: Percentage Change in Roland-Morris Disability Questionnaire (RMDQ) Score
Description: The RMDQ is a self-administered, widely used health status measure for lower back pain (LBP). It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The score of the RMDQ is the total number of items checked - that is from a minimum of 0 (no disability) to a maximum of 24 (maximum disability), where lower scores indicative of better function.
Time Frame: From Baseline to Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0"). Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percentage change in RMDQ score
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 84 | 69
percentage change in RMDQ score | -32.2 (61.81) | -16.4 (41.64)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.103, ANCOVA — The p-value was adjusted using a False Discovery Rate approach (Benjamini-Hochberg); Least Square Mean Difference = -15.9, 95% CI 2-sided [-32.661 to 0.828], Standard Error of Mean 8.47

5. Secondary Outcome: Mobility Evaluation Using Schober's Test
Description: Change in mobility from baseline to Day 5 using Schober's test score.Schober test consists of extending a tape measure on the spinal column, between two posterior superior iliac spines and up to 10 cm above this, with the individual in a neutral position. Then, participant is asked to do anterior flexion of the trunk, then therapist will measure the distance of the marked points, in participants without changes of mobility should increase at least 5 cm. Increases smaller than 5 cm indicate that the test is positive, decreased mobility of the lumbar spine. These data were collected at baseline and at Day 5 and then the change from baseline to Day 5 was calculated for each treatment group.This change from baseline is analyzed by Analysis of covariance(ANCOVA) model with the treatment group as fixed effect and baseline instantaneous pain NRS as continuous covariate.Score range for ITP FIRTECH arm is -2.0 to 6.0 and for no patch control arm is -4.2 to 2.0.
Time Frame: Baseline and Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0"). Number analyzed is the number of participants with data available for analysis at specific timepoint.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
cm
  Baseline: number analyzed (Participants) | 52 | 41
  Baseline | 7.9 (4.52) | 8.1 (4.89)
  Day 5: number analyzed (Participants) | 52 | 40
  Day 5 | 8.7 (5.48) | 8.1 (5.23)
  Change from Baseline: number analyzed (Participants) | 51 | 40
  Change from Baseline | 0.9 (1.44) | -0.1 (1.27)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p < 0.001, ANCOVA — The p-value was adjusted using a False Discovery Rate approach (Benjamini-Hochberg); Least Square Mean Difference = 1.0, 95% CI 2-sided [0.511 to 1.581], Standard Error of Mean 0.27

6. Secondary Outcome: Mobility Evaluation Using Fingertip-to-Floor (FTF) Test
Description: Change in mobility from baseline to Day 5 using FTF test score.Procedure for FTF test follow recommendation of American Psychological Association:participant stood erect on a platform 20-cm high with shoes removed and feet together.Participant was asked to bend forward as far as possible,while maintaining knees,arms,and fingers fully extended.Vertical distance between tip of middle finger and platform is measured with supple tape measure and is expressed in cm.Vertical distance between platform and tip of middle finger is positive when participant did not reach platform and negative when he could go further.These data were collected at baseline and at Day 5 and then change from baseline to Day 5 was calculated for each treatment group.This change from baseline is analyzed by ANCOVA model with treatment group as fixed effect and baseline instantaneous pain NRS as continuous covariate.Score range:ITP FIRTECH arm=-22.0-17.0;no patch control arm=-30.0-13.0.
Time Frame: Baseline and Day 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
cm
  Baseline: number analyzed (Participants) | 87 | 79
  Baseline | 21.0 (17.48) | 18.6 (18.27)
  Day 5: number analyzed (Participants) | 82 | 71
  Day 5 | 17.4 (14.88) | 17.5 (16.41)
  Change from Baseline: number analyzed (Participants) | 80 | 71
  Change from Baseline | -3.5 (6.6) | -1.7 (5.31)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.121, ANCOVA — The p-value was adjusted using a False Discovery Rate approach (Benjamini-Hochberg); Least Square Mean Difference = -1.4, 95% CI 2-sided [-2.976 to 0.250], Standard Error of Mean 0.82

7. Secondary Outcome: Time to Reach Acceptable Pain
Description: Time to reach acceptable pain is defined as the time in hours from baseline subject symptom self-assessment date and time (Day 1 Visit 1, Pain perception) to the first report of post-baseline acceptable pain.
Time Frame: Up to Day 5
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
hours | 9.62 [8.017 to 10.317] | 8.65 [7.250 to 10.533]
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.564, Log Rank — The p-value is adjusted using a False Discovery Rate approach (Benjamini-Hochberg)

8. Secondary Outcome: Time to Reach no Pain
Description: Time to reach no pain was defined as the time (hours) from baseline subject symptom self-assessment date and time (Day 1 Visit
  1, Pain Perception) to the first report of instantaneous pain NRS=0.
Time Frame: Up to Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0"). Overall number analyzed is the number of censored participants with the event.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
hours | NA [NA to NA] — The median and 95% confidence interval (CI) was not estimable as the event did not occur | NA [NA to NA] — The median and 95% CI was not estimable as the event did not occur
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p = 0.289, Log Rank

9. Secondary Outcome: Time Course of PID
Description: NRS is used to assess pain intensity, it is a 11-point scale (0-10) where '0' representing 'no pain' and '10' representing 'worst pain imaginable'. PID was defined as instantaneous pain NRS change from baseline. Instantaneous pain NRS was analyzed from baseline up to Day 5. A negative difference indicates improvement.
Time Frame: Baseline up to Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0"). Number analyzed is the number of participants with data available for analysis at specific timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
units on a scale
  Change from Baseline at Day 1 Evening: number analyzed (Participants) | 82 | 72
  Change from Baseline at Day 1 Evening | -0.8 (1.24) | -0.1 (1.26)
  Change from Baseline at Day 2 Morning: number analyzed (Participants) | 89 | 75
  Change from Baseline at Day 2 Morning | -1.1 (1.55) | -0.6 (1.60)
  Change from Baseline at Day 2 Evening: number analyzed (Participants) | 88 | 71
  Change from Baseline at Day 2 Evening | -1.3 (1.60) | -0.5 (1.76)
  Change from Baseline at Day 3 Morning: number analyzed (Participants) | 85 | 73
  Change from Baseline at Day 3 Morning | -1.6 (1.55) | -0.8 (1.85)
  Change from Baseline at Day 3 Evening: number analyzed (Participants) | 88 | 74
  Change from Baseline at Day 3 Evening | -1.6 (1.53) | -0.9 (1.74)
  Change from Baseline at Day 4 Morning: number analyzed (Participants) | 80 | 69
  Change from Baseline at Day 4 Morning | -1.8 (1.44) | -0.9 (1.91)
  Change from Baseline at Day 4 Evening: number analyzed (Participants) | 92 | 76
  Change from Baseline at Day 4 Evening | -1.8 (1.56) | -1.0 (1.99)
  Change from Baseline at Day 5 Morning: number analyzed (Participants) | 67 | 56
  Change from Baseline at Day 5 Morning | -1.6 (1.58) | -1.0 (2.20)
  Change from Baseline at Day 5: number analyzed (Participants) | 88 | 75
  Change from Baseline at Day 5 | -2.1 (1.64) | -1.4 (1.85)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 1 Evening; Test type: Superiority; p = 0.001, Satterthwaite t-test
Statistical Analysis 2: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 2 Morning; Test type: Superiority; p = 0.035, Satterthwaite t-test
Statistical Analysis 3: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 2 Evening; Test type: Superiority; p = 0.004, Satterthwaite t-test
Statistical Analysis 4: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 3 Morning; Test type: Superiority; p = 0.007, Satterthwaite t-test
Statistical Analysis 5: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 3 Evening; Test type: Superiority; p = 0.005, Satterthwaite t-test
Statistical Analysis 6: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 4 Morning; Test type: Superiority; p = 0.001, Satterthwaite t-test
Statistical Analysis 7: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 4 Evening; Test type: Superiority; p = 0.007, Satterthwaite t-test
Statistical Analysis 8: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 5 Morning; Test type: Superiority; p = 0.096, Satterthwaite t-test
Statistical Analysis 9: Comparison: ITP FIRTECH vs No Patch Control Arm; Change from Baseline at Day 5; Test type: Superiority; p = 0.015, Satterthwaite t-test

10. Secondary Outcome: Time Course of Pain Relief
Description: Pain relief is assessed using a verbal rating scale (VRS), where 0 = none and 4 = complete in response to a pain relief question.
Time Frame: Baseline up to Day 5
Population: Full Analysis Set population was defined as all participants randomized that had the NRS evaluation done at baseline and that were not using any rescue medication starting from randomization to Day 5 Visit 2 or starting before the study and still ongoing at randomization with the exclusion of participants without any pain at baseline (i.e. baseline instantaneous pain NRS score equal to "0"). Number analyzed is the number of participants with data available at specific timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
units on a scale
  Day 1 Evening: number analyzed (Participants) | 82 | 72
  Day 1 Evening | 0.8 (0.86) | 0.3 (0.61)
  Day 2 Morning: number analyzed (Participants) | 89 | 75
  Day 2 Morning | 1.2 (0.97) | 0.7 (1.01)
  Day 2 Evening: number analyzed (Participants) | 88 | 71
  Day 2 Evening | 1.2 (0.92) | 0.7 (0.97)
  Day 3 Morning: number analyzed (Participants) | 85 | 73
  Day 3 Morning | 1.4 (1.03) | 0.7 (0.91)
  Day 3 Evening: number analyzed (Participants) | 88 | 74
  Day 3 Evening | 1.4 (0.98) | 0.7 (1.02)
  Day 4 Morning: number analyzed (Participants) | 80 | 69
  Day 4 Morning | 1.6 (1.11) | 0.8 (1.07)
  Day 4 Evening: number analyzed (Participants) | 92 | 76
  Day 4 Evening | 1.6 (1.16) | 0.9 (1.17)
  Day 5 Morning: number analyzed (Participants) | 67 | 56
  Day 5 Morning | 1.6 (1.22) | 1.1 (1.37)
  Day 5: number analyzed (Participants) | 88 | 75
  Day 5 | 1.9 (1.21) | 0.9 (1.32)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 1 Evening; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 2: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 2 Morning; Test type: Superiority; p = 0.001, Satterthwaite t-test
Statistical Analysis 3: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 2 Evening; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 4: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 3 Morning; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 5: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 3 Evening; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 6: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 4 Morning; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 7: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 4 Evening; Test type: Superiority; p < 0.001, Satterthwaite t-test
Statistical Analysis 8: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 5 Morning; Test type: Superiority; p = 0.024, Satterthwaite t-test
Statistical Analysis 9: Comparison: ITP FIRTECH vs No Patch Control Arm; VRS: Day 5; Test type: Superiority; p < 0.001, Satterthwaite t-test

11. Secondary Outcome: Normalized Sum of Pain Relief
Description: Total pain relief (TOTPAR) is calculated by multiplying the pain relief score at each post-dose time point by the duration (in hours) since the preceding time point. The Normalized Sum of Pain Relief (TOTPAR0- 5) is to be calculated as the Total Pain Relief divided by the total duration time. Higher scores indicate more pain relief. The score range is from 0.0 to 3.5 for both the arms.
Time Frame: Baseline up to Day 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITP FIRTECH | No Patch Control Arm
Number analyzed (Participants) | 97 | 84
units on a scale | 1.46 (0.834) | 0.78 (0.842)
Statistical Analysis 1: Comparison: ITP FIRTECH vs No Patch Control Arm; Test type: Superiority; p < 0.001, ANCOVA; Least Square Mean Difference = 0.7, 95% CI 2-sided [0.415 to 0.903], Standard Error of Mean 0.12

ADVERSE EVENTS:
Time Frame: Day 1 to Day 6
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events is mentioned for Safety Population. Safety population was defined as all participants randomized into the study and, if randomized to the "patch" arm, had the device installed.
Arm/Group | ITP FIRTECH | No Patch Control Arm
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/107
Other Adverse Events (participants affected / at risk) | 18/114 | 7/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITP FIRTECH (N=114) | No Patch Control Arm (N=107)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application Site Erythema (General disorders) | 2 (2) | 0 (0)
Application Site Irritation (General disorders) | 1 (1) | 0 (0)
Application Site Pain (General disorders) | 2 (2) | 0 (0)
Application Site Paraesthesia (General disorders) | 1 (1) | 0 (0)
Application Site Pruritus (General disorders) | 7 (8) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT05137041/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT05137041/SAP_001.pdf